CLINICAL TRIAL: NCT04481217
Title: The Mediating Role of Dissociative Symptoms and Early Maladaptive Schemas in the Relationship Between Childhood Trauma and Auditory Hallucinations in Schizophrenia
Brief Title: Cognitive Factors Mediating the Relationship Between Childhood Trauma and Auditory Hallucinations in Schizophrenia
Acronym: HADITRYOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC20.055; 2020-A00452-37 (Other: ID RCB)
Record Dates: First submitted 2020-05-22; First posted 2020-07-22 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Schizophrenia
Keywords: schizophrenia; auditory verbal hallucinations; early maladaptive schemas; dissociative symptoms; childhood traumas; mediation modeling
MeSH Terms: conditions — Schizophrenia; Hallucinations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Schizophrenia (Experimental): Patients included will be diagnosed with schizophrenia or schizoaffective disorder, and experience AVH at the time of the inclusion (n= 350). All will be inpatients.
  Interventions: Other: Self-questionnaires battery; Other: Socio-demographic screening

INTERVENTIONS:
Other: Self-questionnaires battery — * Childhood trauma questionnaire (Bernstein, Ahluvalia, Pogge, & Handelsman, 1997; Bernstein et al., 2003)
  * The Young schema questionnaire short form (SQ-SF ; Cottraux & Black, 2006; Young, 1998).
  * Dissociative experiences scale (Laroi et al., 2013).
  * Launay-Slade hallucination scale (Bentall & Slade, 1985; Launay & Slade, 1981)
  * Cardiff Anomalous Perceptions Scale (Bell et al., 2006)
Other: Socio-demographic screening — age; gender; education; highest diploma; job; marital status; living place

SUMMARY:
BACKGROUND It is demonstrated that strong associations between trauma suffered in childhood and having schizophrenia, and more specifically to experience acoustic-verbal hallucinations (AVH). A second generation of research is currently examining the cognitive and affective processes likely to play a mediating role in this association. These mediators appear to include early maladaptive personality patterns and dissociative experiences. Although these factors have most often been explored separately, recent research indicates that they could be associated, and thus contribute to AVH. More specifically, another study has shown that the association between childhood trauma and predisposition to AVH is not direct but depends on cognitive factors including the impact of violence suffered during childhood on early maladaptive schemas and dissociation. However, this study was carried out on a non-clinical sample of subjects with a predisposition to AVH.

OBJECTIVES: testing a structural model of AVH, childhood trauma, early maladaptive schemas and dissociative symptoms in large multicentric sample of inpatients diagnosed with schizophrenia and AVH (n=350). Secondary objectives are (i) test in the model the role of all the early patterns described by Jeffrey Young instead of targeting only the schemes that are part of the model tested in previous study as the one by Bortolon and colleagues, (ii) compare the quality of the adjustment of the confirmatory model to the quality of the adjustment of the exploratory model.

METHODS: one single visit in which subjects will receive self-reported questionnaires (Childhood trauma questionnaire, The Young schema questionnaire short form, Dissociative experiences scale, Launay-Slade hallucination scale and Cardiff Anomalous Perceptions Scale.

ANALYSES: Structural equation model performed additional analysis using Partial Least Squares Structural Equation Modelling. The primary endpoint corresponds to significant associations between the variables. The quality of the model will be assessed using a fit quality measure. The secondary endpoints are significant associations between the different variables (p <0.05) and the model quality assessed with a quality measure of the fit.

MAIN HYPOTHESIS: the association between childhood trauma and predisposition to AVH is not direct, but depends on the impact of violence suffered during childhood on early maladaptive schemas and dissociative symptoms in patients with schizophrenia.

DETAILED DESCRIPTION:
BACKGROUND A first generation of research has demonstrated strong associations between trauma suffered in childhood (physical, psychological and sexual violence) and having schizophrenia, and more specifically to experience "hearing voices" (acoustic-verbal hallucinations, AVH).

A second generation of research is currently examining the cognitive and affective processes likely to play a mediating role in this association. These mediators appear to include early maladaptive personality patterns and dissociative experiences. Although these factors have most often been explored separately, recent research indicates that they could be associated, and thus contribute to AVH. More specifically, another study has shown that the association between childhood trauma and predisposition to AVH is not direct but depends on cognitive factors including the impact of violence suffered during childhood on early maladaptive schemas (for example, interpersonal functioning centred on "subjugation", "abandonment", "vulnerability") and dissociation. However, this study was carried out on a non-clinical sample of subjects with a predisposition to AVH OBJECTIVES Here, aim is at testing a structural model of AVH, childhood trauma, early maladaptive schemas and dissociative symptoms in large sample of patients diagnosed with schizophrenia and AVH (n=350).

Secondary objectives are (i) to carry out exploratory analyzes which will allow investigators to test in the model the role of all the early patterns described by Jeffrey Young instead of targeting only the schemes that are part of the model tested in previous study as the one by Bortolon and colleagues, (ii) compare the quality of the adjustment of the confirmatory model to the quality of the adjustment of the exploratory model.

METHODS

A cross-sectional, multicenter design (3 centres) will be performed. Patients included will be diagnosed with schizophrenia or schizoaffective disorder, and experience AVH at the time of the inclusion (n= 350). All will be inpatients. The study consists of one single visit in which the subjects will receive all the self-reported questionnaires to be completed:

1. General information sheet (socio-demographic and clinical data)
2. Questionnaire on traumatic childhood experiences: Childhood trauma questionnaire
3. Questionnaire on early maladaptive schemas: The Young schema questionnaire short form
4. Questionnaire about dissociative experiences: Dissociative experiences scale
5. Questionnaire on hallucinations: Launay - Slade hallucination scale and Cardiff Anomalous Perceptions Scale.

All questionnaires have been validated in French. ANALYSES Structural equation model performed additional analysis using Partial Least Squares Structural Equation Modelling (PLS-SEM).

The primary endpoint corresponds to significant associations (significance threshold <0.05) between the variables as in the model described by Bortolon and colleagues. The quality of the model (both measurement and structural model) will be assessed using a fit quality measure.

The secondary endpoints are significant associations between the different variables (p <0.05) and the model quality assessed with a quality measure of the fit.

HYPOTHESES It's hypothesized that the association between childhood trauma and predisposition to AVH is not direct, but depends on the impact of violence suffered during childhood on early maladaptive schemas (for example, interpersonal functioning centred on "subjugation", "abandonment", "vulnerability") and dissociative symptoms in patients with schizophrenia.

ELIGIBILITY:
Inclusion criteria:

* Schizophrenia or schizo-affective disorder
* Auditory hallucinations
* Fluent in French
* Gave informed consent

Exclusion Criteria:

* Agitation or suicide risk
* Involuntary Hospitalization
* Neurologic condition
* No informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350 (Estimated)
Dates: Start 2020-09-04 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Auditory hallucinations measured by the Launay-Slade Hallucination Scale | Baseline
  The auditory hallucinations measured by the Launay-Slade Hallucination Scale, which is a self-report scale developed to measure predisposition to hallucinations.
  Three items were designed to measure verbal hallucinations, which are measured using a 5-point Likert scale, from 0 to 4 (0 = "definitely does not apply to me," 1 = "possibly does not apply to me," 2 = "unsure," 3 = "possibly applies to me," and 4 = "definitely applies to me").

SECONDARY OUTCOMES:
Defensive dissociation assessed by the Dissociative experiences scale (DES) | Baseline
  Defensive dissociation assessed by the Dissociative experiences scale (DES). The DES is a 28-item developed to measure dissociative experiences. Respondents are asked to rate how often they experienced each of the 28 described situation compared to other people. The scale was composed of 11 boxes that the participants had to tick (from "much less than others" to "much more than others").
Early maladaptive schema "Abandonment", which is measured by the young schema questionnaire short form (SQ-SF) | Baseline
  The early maladaptive schema "Abandonment", which is measured by the young schema questionnaire short form (SQ-SF). The SQ-SF is a 75-item, self-report inventory designed to measure 15 EMS proposed by Young. Each item is rated on a 6-point scale (from 1 = "completely untrue of me" to 6 = "describes me perfectly"). Higher scores indicate a greater presence of a maladaptive schema for the respondent.
The early maladaptive schema "Self-sacrifice", which is measured by the young schema questionnaire short form (SQ-SF) | Baseline
  The early maladaptive schema "Self-sacrifice", which is measured by the young schema questionnaire short form (SQ-SF). The SQ-SF is a 75-item, self-report inventory designed to measure 15 EMS proposed by Young. Each item is rated on a 6-point scale (from 1 = "completely untrue of me" to 6 = "describes me perfectly"). Higher scores indicate a greater presence of a maladaptive schema for the respondent.
The early maladaptive schema "Vulnerability", which is measured by the young schema questionnaire short form (SQ-SF) | Baseline
  The early maladaptive schema "Vulnerability", which is measured by the young schema questionnaire short form (SQ-SF). The SQ-SF is a 75-item, self-report inventory designed to measure 15 EMS proposed by Young. Each item is rated on a 6-point scale (from 1 = "completely untrue of me" to 6 = "describes me perfectly"). Higher scores indicate a greater presence of a maladaptive schema for the respondent.
The early maladaptive schema "Subjugation", which is measured by the young schema questionnaire short form (SQ-SF) | Baseline
  The early maladaptive schema "Subjugation", which is measured by the young schema questionnaire short form (SQ-SF). The SQ-SF is a 75-item, self-report inventory designed to measure 15 EMS proposed by Young. Each item is rated on a 6-point scale (from 1 = "completely untrue of me" to 6 = "describes me perfectly"). Higher scores indicate a greater presence of a maladaptive schema for the respondent.

CONTACTS AND LOCATIONS:
Overall Officials: Clément DONDE, Principal Investigator — CHU Grenoble Alpes
Locations (2):
- France (2):
  - Grenoble University Hospital, La Tronche
  - Chu St Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daalman K, Diederen KM, Derks EM, van Lutterveld R, Kahn RS, Sommer IE. Childhood trauma and auditory verbal hallucinations. Psychol Med. 2012 Dec;42(12):2475-84. doi: 10.1017/S0033291712000761. Epub 2012 Apr 16. PMID 22716897
- [Background] Varese F, Smeets F, Drukker M, Lieverse R, Lataster T, Viechtbauer W, Read J, van Os J, Bentall RP. Childhood adversities increase the risk of psychosis: a meta-analysis of patient-control, prospective- and cross-sectional cohort studies. Schizophr Bull. 2012 Jun;38(4):661-71. doi: 10.1093/schbul/sbs050. Epub 2012 Mar 29. PMID 22461484
- [Background] Williams J, Bucci S, Berry K, Varese F. Psychological mediators of the association between childhood adversities and psychosis: A systematic review. Clin Psychol Rev. 2018 Nov;65:175-196. doi: 10.1016/j.cpr.2018.05.009. Epub 2018 Jun 2. PMID 30243100
- [Background] Bortolon C, Seille J, Raffard S. Exploration of trauma, dissociation, maladaptive schemas and auditory hallucinations in a French sample. Cogn Neuropsychiatry. 2017 Nov;22(6):468-485. doi: 10.1080/13546805.2017.1387524. Epub 2017 Oct 12. PMID 29023198
- [Background] Evans GJ, Reid G, Preston P, Palmier-Claus J, Sellwood W. Trauma and psychosis: The mediating role of self-concept clarity and dissociation. Psychiatry Res. 2015 Aug 30;228(3):626-32. doi: 10.1016/j.psychres.2015.04.053. Epub 2015 Jun 11. PMID 26099655
- [Background] Bell V. A community of one: social cognition and auditory verbal hallucinations. PLoS Biol. 2013 Dec;11(12):e1001723. doi: 10.1371/journal.pbio.1001723. Epub 2013 Dec 3. PMID 24311984
- [Background] Bentall RP, Slade PD. Reality testing and auditory hallucinations: a signal detection analysis. Br J Clin Psychol. 1985 Sep;24 ( Pt 3):159-69. doi: 10.1111/j.2044-8260.1985.tb01331.x. PMID 4052663
- [Background] Laroi F, Marczewski P, Van der Linden M. Further evidence of the multi-dimensionality of hallucinatory predisposition: factor structure of a modified version of the Launay-Slade Hallucinations Scale in a normal sample. Eur Psychiatry. 2004 Feb;19(1):15-20. doi: 10.1016/S0924-9338(03)00028-2. PMID 14969776
- [Background] Cottraux J, & Blackburn IM. Psychothérapies cognitives des troubles de la personnalité. NPG Neurologie-Psychiatrie-Gériatrie. 2007; 7(37), 41.
- [Background] Larøi F, Billieux J, Defeldre A-C, Ceschi, G, Van der Linden M. Factorial structure and psychometric properties of the French adaptation of the Dissociative Experiences Scale (DES) in non-clinical participants. Revue Européenne de Psychologie Appliquée/European Review of Applied Psychology. 2013; 63(4): 203-208.
- [Background] Launay G, Slade P. The measurement of hallucinatory predisposition in male and female prisoners. Personality and Individual Differences. 1981; 2(3): 221-234.
- [Background] Mauchand P, Lachenal-Chevallet K, Cottraux J. [Empirical validation of the Young Schema Questionnaire-Short Form (YSQ-S2) in borderline personality disorder and control subjects]. Encephale. 2011 Apr;37(2):138-43. doi: 10.1016/j.encep.2010.04.014. Epub 2010 Jul 3. French. PMID 21482232
- [Background] Briere J, Scott C. Assessment of trauma symptoms in eating-disordered populations. Eat Disord. 2007 Jul-Sep;15(4):347-58. doi: 10.1080/10640260701454360. PMID 17710571
- [Background] Darves-Bornoz JM, Degiovanni A, Gaillard P. Validation of a French version of the Dissociative Experiences Scale in a rape-victim population. Can J Psychiatry. 1999 Apr;44(3):271-5. doi: 10.1177/070674379904400308. PMID 10225129
- [Background] Garrison JR, Moseley P, Alderson-Day B, Smailes D, Fernyhough C, Simons JS. Testing continuum models of psychosis: No reduction in source monitoring ability in healthy individuals prone to auditory hallucinations. Cortex. 2017 Jun;91:197-207. doi: 10.1016/j.cortex.2016.11.011. Epub 2016 Nov 22. PMID 27964941
- [Background] Johns LC, Kompus K, Connell M, Humpston C, Lincoln TM, Longden E, Preti A, Alderson-Day B, Badcock JC, Cella M, Fernyhough C, McCarthy-Jones S, Peters E, Raballo A, Scott J, Siddi S, Sommer IE, Laroi F. Auditory verbal hallucinations in persons with and without a need for care. Schizophr Bull. 2014 Jul;40 Suppl 4(Suppl 4):S255-64. doi: 10.1093/schbul/sbu005. PMID 24936085
- [Background] Perona-Garcelan S, Carrascoso-Lopez F, Garcia-Montes JM, Ductor-Recuerda MJ, Lopez Jimenez AM, Vallina-Fernandez O, Perez-Alvarez M, Gomez-Gomez MT. Dissociative experiences as mediators between childhood trauma and auditory hallucinations. J Trauma Stress. 2012 Jun;25(3):323-9. doi: 10.1002/jts.21693. Epub 2012 May 15. PMID 22589015
- [Background] Perona-Garcelan S, Garcia-Montes JM, Cuevas-Yust C, Perez-Alvarez M, Ductor-Recuerda MJ, Salas-Azcona R, Gomez-Gomez MT. A preliminary exploration of trauma, dissociation, and positive psychotic symptoms in a Spanish sample. J Trauma Dissociation. 2010;11(3):284-92. doi: 10.1080/15299731003786462. PMID 20603763
- [Background] Pilton M, Varese F, Berry K, Bucci S. The relationship between dissociation and voices: A systematic literature review and meta-analysis. Clin Psychol Rev. 2015 Aug;40:138-55. doi: 10.1016/j.cpr.2015.06.004. Epub 2015 Jun 16. PMID 26117061
- [Background] Wright DB, Loftus EF. Measuring dissociation: comparison of alternative forms of the dissociative experiences scale. Am J Psychol. 1999 Winter;112(4):497-519. PMID 10696264
- [Background] Wright MO, Crawford E, Del Castillo D. Childhood emotional maltreatment and later psychological distress among college students: the mediating role of maladaptive schemas. Child Abuse Negl. 2009 Jan;33(1):59-68. doi: 10.1016/j.chiabu.2008.12.007. Epub 2009 Jan 23. PMID 19167067
- [Background] Young JE. Cognitive therapy for personality disorders : A schema-focused approach. Professional Resource Press/Professional Resource Exchange. 1999.
- [Background] Young JE, Brown G. Young schema questionnaire short form. New York: Cognitive Therapy Centre. 1998.
- [Background] Young JE, Klosko, JS, Weishaar, ME. Schema therapy : A practitioner's guide. 2005.
- [Background] Hair Jr JF, Hult GTM, Ringle C, Sarstedt M. A primer on partial least squares structural equation modeling (PLS-SEM). Sage publications. 2016.
- [Background] First MB, Spitzer RL, Gibbon M, Williams JB, et al. Structured clinical interview for DSM-IV axis I disorders. New York: New York State Psychiatric Institute. 1995.
- [Background] Battle DE. Diagnostic and Statistical Manual of Mental Disorders (DSM). Codas. 2013;25(2):191-2. doi: 10.1590/s2317-17822013000200017. No abstract available. PMID 24413388
- [Background] Bernstein DP, Ahluvalia T, Pogge D, Handelsman L. Validity of the Childhood Trauma Questionnaire in an adolescent psychiatric population. J Am Acad Child Adolesc Psychiatry. 1997 Mar;36(3):340-8. doi: 10.1097/00004583-199703000-00012. PMID 9055514
- [Background] Bernstein DP, Stein JA, Newcomb MD, Walker E, Pogge D, Ahluvalia T, Stokes J, Handelsman L, Medrano M, Desmond D, Zule W. Development and validation of a brief screening version of the Childhood Trauma Questionnaire. Child Abuse Negl. 2003 Feb;27(2):169-90. doi: 10.1016/s0145-2134(02)00541-0. PMID 12615092